CLINICAL TRIAL: NCT01724359
Title: An Open-label Prospective Trial to Explore the Tolerability, Safety and Efficacy of Flexibly Dosed Paliperidone ER in Subjects With Schizophrenia
Brief Title: Tolerability, Safety and Efficacy of Flexibly Dosed Paliperidone ER in Patients With Schizophrenia
Acronym: PERFLEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017413; R076477SCH3029 (Other: Janssen-Cilag Colombia); R076477SCH3036 (Other: Janssen-Cilag Argentina)
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone extended-release (ER); Antipsychotic agents
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone ER (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — The recommended Paliperidone extended-release (ER) dose will be 6 mg/day. Some patients may benefit from higher or lower doses, in the range of 3 to 12 mg/day. Paliperidone ER will be administered orally once daily. Adjustment of the dosage will be done at the investigator's discretion.

SUMMARY:
The purpose of this study is to evaluate efficacy, safety and tolerability of flexible, once-daily doses of paliperidone extended-release (ER) in patients with schizophrenia from Argentina and Colombia that previously failed treatment with other antipsychotic agents.

DETAILED DESCRIPTION:
This is a single arm (one group of patients), open-label (all people know the identity of the intervention) multicenter 6-month study. Throughout the study flexible dosing of paliperidone ER in a range of 3 to 12 mg/day may be used. Flexible dosing will allow investigators to adjust the dosage of each patient based on the individual needs. Patients will receive 3, 6, 9 or 12 mg of paliperidone ER once daily for 6 months. The tablets will be taken orally. Adjustment of the dosage will be done at the investigator's discretion, based on the individual patient's clinical response and tolerability to the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the criteria for schizophrenia
* Patient is previously non-acute and has been given an adequate dose of an appropriate oral antipsychotic for an adequate period of time prior to enrollment, but previous treatment is considered unsuccessful due to one or more of the following reasons: lack of efficacy, lack of tolerability or safety, lack of compliance and/or other reasons to switch to another antipsychotic medication
* Patient is healthy on the basis of a physical examination and vital signs at screening
* Women must be postmenopausal for at least 1 year, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry and throughout the study

Exclusion Criteria:

* Patients on clozapine, any conventional depot neuroleptic or risperidone long-acting injections during the last 3 months
* Patients with serious unstable medical condition, including known clinically relevant laboratory abnormalities
* Patients with history or current symptoms of tardive dyskinesia and neuroleptic malignant syndrome
* Patients judged to be at high risk for adverse events, violence, or self-harm
* Patients with known hypersensitivity to paliperidone ER or to risperidone
* Patients with a current use or known history (over the past 6 months) of substance dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. Clinical Trial, Study Director — Janssen-Cilag, S.A.
Locations (5):
- Argentina (2):
  - Buenos Aires
  - Rosario
- Colombia (3):
  - Bogotá
  - Cali
  - Medellín

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who received paliperidone extended-release (ER) at least once and provide at least 1 post baseline efficacy measurement will be included in the intent-to-treat (ITT) analysis set for efficacy. Patients who received paliperidone ER at least once and provide any post-baseline information will be included in the ITT analysis set for safety.
Groups:
- Paliperidone Extended-release (ER): The recommended Paliperidone ER dose is 6 mg/day. Some patients may benefit from higher or lower doses, in the range of 3 to 12 mg/day. Paliperidone ER will be administered orally once daily.
Period: Overall Study
Arm/Group | Paliperidone Extended-release (ER)
Started | 95
Completed | 64
Not Completed | 31
Not completed — Adverse Event | 10
Not completed — Death | 1
Not completed — Other | 20

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 95
Age Continuous [Mean (Standard Deviation); unit: years] | 35.86 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 54
Region of Enrollment [Number; unit: participants]
  Argentina | 37
  Colombia | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Positive and Negative Syndrome Scale (PANSS) Score
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 70
scores on a scale
  Baseline (n= 70) | 83.99 (22.16)
  Week 26 (n= 70) | 53.70 (18.82)

2. Secondary Outcome: Change From Baseline in Total Positive and Negative Syndrome Scale (PANSS) - Positive Subscale Score
Description: The PANSS Positive Subscale assesses seven positive-symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 70
scores on a scale
  Baseline (n= 70) | 18.53 (7.30)
  Week 26 (n= 70) | 11.16 (4.95)

3. Secondary Outcome: Change From Baseline in Total Positive and Negative Syndrome Scale (PANSS) - Negative Subscale Score
Description: The PANSS Negative Subscale assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 70
scores on a scale
  Baseline (n= 70) | 23.69 (6.42)
  Week 26 (n= 70) | 14.64 (5.24)

4. Secondary Outcome: Change From Baseline in Total Positive and Negative Syndrome Scale (PANSS) - General Psychopathology Subscale Score
Description: The PANSS General Psychopathology Subscale Score assesses 16 general psychopathology symptoms. The symptoms are rated on a 7-point scale, with a range of 16 (absent) to 112 (extreme psychopathology).
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 70
scores on a scale
  Baseline (n= 70) | 41.77 (11.39)
  Week 26 (n= 70) | 27.90 (10.34)

5. Secondary Outcome: Clinical Global Impression-Severity (CGIS)
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients". Higher scores indicate worsening.
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Number; unit: participants
Groups:
- Patients at Baseline: Paliperidone Extended-release (ER); Patients at Week 26: Paliperidone Extended-release (ER): The recommended Paliperidone ER dose is 6 mg/day. Some patients may benefit from higher or lower doses, in the range of 3 to 12 mg/day. Paliperidone ER will be administered orally once daily.
Arm/Group | Patients at Baseline: Paliperidone Extended-release (ER) | Patients at Week 26: Paliperidone Extended-release (ER)
Number analyzed (Participants) | 95 | 83
participants
  Normal, not at all ill | 2 | 9
  Borderline mentally ill | 3 | 21
  Mildly ill | 14 | 26
  Moderately ill | 39 | 20
  Markedly ill | 26 | 5
  Severely ill | 10 | 2
  Among the most extremely ill | 1 | 0

6. Secondary Outcome: Personal and Social Performance (PSP) Scale
Description: This PSP assesses the degree of a patient's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (i, absent to vi, very severe) in each of the 4 domains. Based on the four domains there will be one total score. Patients with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; =< 30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 95
scores on a scale
  Baseline (n= 95) | 52.06 (15.27)
  Week 26 (n= 78) | 68.24 (15.91)

7. Secondary Outcome: Health Status as Measured by Self-rated Health Status Survey SF-36
Description: The SF-36 is designed to examine a person's perceived health status. The SF-36 includes one multi-item scale measuring eight health concepts: vitality, physical functioning, bodily pain, general health perceptions, physical role-, emotional role-, social role functioning, and mental health. Answers to each question are scored and summed to produce raw scale scores for each health concept which are then transformed to a 0 - 100 scale, a high score defining a more favorable health state. An aggregate summary measure is calculated by averaging the scores from the eight health concepts.
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 95
scores on a scale
  Baseline (n= 95) | 56.39 (18.14)
  Week 26 (n= 86) | 67.02 (21.56)

8. Secondary Outcome: Sleep Evaluation Scale
Description: This self-administered scale rates the quality of sleep. Patients will indicate on an 11-point scale how well they have slept in the previous 7 days, from 0 (very badly) to 10 (very well).
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 71
scores on a scale
  Baseline (n= 71) | 6.80 (2.69)
  Week 26 (n= 71) | 7.66 (2.52)

9. Secondary Outcome: Daytime Drowsiness Evaluation Scale
Description: This self-administered scale rates the daytime drowsiness. Patients will indicate on an 11-point scale how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 10 (all the time).
Time Frame: Baseline, Week 26
Population: All participants of the intent-to-treat analysis set for efficacy with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 71
scores on a scale
  Baseline (n= 71) | 4.68 (3.21)
  Week 26 (n= 71) | 2.58 (2.93)

ADVERSE EVENTS:
Arm/Group | Paliperidone Extended-release (ER)
Serious Adverse Events (participants affected / at risk) | 7/95
Other Adverse Events (participants affected / at risk) | 39/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended-release (ER) (N=95)
Psychotic episode (Psychiatric disorders) | 3
Clinical deterioration (General disorders) | 1
Appendicitis (Gastrointestinal disorders) | 1
Major depressive disorder (Psychiatric disorders) | 1
Worsening of the psychiatric condition with aggressive behavior (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended-release (ER) (N=95)
Akathisia (Nervous system disorders) | 22
Insomnia (Psychiatric disorders) | 24
Parkinsonism (Nervous system disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less